CLINICAL TRIAL: NCT07336238
Title: A Phase 2a Study of Group Retreat Psilocybin Therapy for Cancer-Related Anxiety and Depression
Brief Title: Group Retreat Psilocybin Therapy for the Treatment of Anxiety and Depression in Patients With Metastatic Solid Tumors or Incurable Hematologic Malignancies
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Healing Hearts, Changing Minds, Inc. (Unknown); Psilo Scientific Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1126153; NCI-2025-09712 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Depression; Hematopoietic and Lymphatic System Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasm Metastasis | interventions — Psychotherapy; Therapeutics; Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (psilocybin therapy) (Experimental): Patients attend group preparation therapy sessions on days -14 (virtual), -7 (virtual) and -1 (in person), and also attend an individual preparation therapy session on day -1 (in person). Patients receive psilocybin orally (PO) on day 0. Patients may receive an additional "booster" dose 60-90 minutes after the initial dose based on the physician's clinical judgement. Patients attend group integration therapy sessions on days 1 (in person), 8 (virtual), 15 (virtual), and 22 (virtual), and attend individual integration therapy sessions on days 1 (in person) and 8 (virtual).
  Interventions: Behavioral: Psychotherapy; Drug: Psilocybin; Other: Survey Administration

INTERVENTIONS:
Behavioral: Psychotherapy — Attend therapy sessions
  Other Names: therapy; talk therapy
Drug: Psilocybin — Given PO
  Other Names: psilocybine
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II trial tests the safety, side effects and how well group retreat psilocybin therapy works for the treatment of anxiety and depression in patients with solid tumors that have spread from where they first started (primary site) to other places in the body (metastatic) or with hematologic cancers for which no treatment is currently available (incurable). For patients with metastatic, incurable cancer, unrelieved anxiety and existential distress can cause profound suffering. Psilocybin therapy can relieve anxiety and existential distress by disrupting patterns of thinking that contribute to anxiety and depression. Psilocybin is a substance being studied in the treatment of anxiety or depression in patients with cancer. In this study, a pharmaceutical grade of psilocybin will be used that has been approved by the FDA for research, provided by Filament Health. Psilocybin acts on the brain by resetting the brain's activity and increasing connections between brain regions, particularly those involved in mood regulation and self-perception. In this study psilocybin is combined with structured discussions and reflections that enable patients to have new insights about their situation. In a prior study, group retreat psilocybin therapy was proven to be safe and this study tests a refined dosing regimen for symptoms of anxiety and depression in patients with metastatic solid tumors or incurable hematologic malignancies.

DETAILED DESCRIPTION:
OUTLINE:

Patients attend group preparation therapy sessions on days -14 (virtual), -7 (virtual) and -1 (in person), and also attend an individual preparation therapy session on day -1 (in person). Patients receive psilocybin orally (PO) on day 0. Patients may receive an additional "booster" dose 60-90 minutes after the initial dose based on their subjective report combined with the physician's clinical judgement. Patients attend group integration therapy sessions on days 1 (in person), 8 (virtual), 15 (virtual), and 22 (virtual), and attend individual integration therapy sessions on days 1 (in person) and 8 (virtual).

After completion of study treatment, patients are followed up at 8, 12, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of metastatic solid tumor, or incurable hematologic malignancy that has been accepted by a physician in a medical record
* Measurable disease is not required
* Previous treatment with chemotherapy: There are no minimum or maximum prior lines of chemotherapy
* 18-85 years of age
* Required performance status, including the appropriate scale. Eastern Cooperative Oncology Group (ECOG) 0-2
* Hematocrit > 20
* Platelets (plt) > 20K
* Liver function tests 1.5 x normal
* Creatinine 1.5 x normal
* Subjects of childbearing potential must be willing to use an effective contraceptive method from study enrollment until at least 1 month after receiving the investigational agent(s)
* Must be at least 4 weeks after surgery or radiotherapy at study entry, but can be receiving oral or intravenous (IV) chemotherapy if those schedules can be adjusted around the medication session date
* Motivated to participate in a group study and able in the research team's judgment to participate in the small group effectively
* On pre-enrollment screening tests, they will have clinically significant anxiety or depressive symptoms as defined by a score of 11 or greater on the Hospital and Anxiety Depression Scale-Anxiety (HADS)-total
* English speaking - able to understand the process of consent and the risk and benefits associated with the study, and able to give written informed consent. This is a pilot study, and if future larger studies are designed, consideration will be given for non-english-speaking subjects
* Must be willing to sign a medical release for the investigators to communicate directly with their treating clinicians (mental health professional or oncologist) and doctors to confirm a medication and/or medical history
* Must provide at least one adult who is in contact with the participant at least once a day when the participant is at home who is able to verbally monitor participant-reported changes in the behavior and able to notify research staff of behavior changes that may require research staff assessment
* Must provide a review of any selective serotonin reuptake inhibitor (SSRI) use
* Must avoid taking any psychiatric medications or starting a new psychiatric medication during the study. Should participant's doctor recommend starting a new psychiatric medication, participant will be required to notify the study team and the subject would withdraw from the study. (Use of as needed [prn] benzodiazepines is allowed but high dose chronic benzodiazepine use must be reviewed by the principal investigator [PI]. Use of prn gabapentoids is allowed but high dose chronic gabapentoid use must be reviewed by the PI.)
* Must provide a contact (relative, spouse, close friend, or other caregiver) who is willing and able to be reached by the research team in the event that the participant becomes suicidal
* If the potential participant is of childbearing potential, they must have a negative pregnancy test at baseline and prior to the medication dosing session, and must agree to use highly effective birth control. Highly effective birth control is defined as birth control methods, alone or in combination, that result in a low failure rate (i.e., less than 1 percent per year, which does NOT include condoms or abstinence
* Are willing to commit to preparation sessions, medication dosing sessions, integration sessions, to complete evaluation instruments and commit to be contacted for all necessary telephone contacts

Exclusion Criteria:

* Brain metastases that have not been treated
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy, breastfeeding, or expecting to conceive or father children for the duration of the trial through 30 days after receipt of investigational agent(s)
* Personal or immediate family history of schizophrenia, bipolar affective disorder, delusion disorder, paranoid disorder, or schizoaffective disorder
* Suicidal ideation with a Columbia-Suicide Severity Rating Scale (C-SSRS) measurement of 'low risk' or no risk
* Current substance abuse disorder (although prospective subjects will not be excluded for reasonable alcohol use that does not meet criteria for alcohol use disorder or marijuana use that does not meet criteria for substance use disorder)
* Unstable neurological or medical condition; history of seizure, chronic/severe headaches
* Any use of psychedelic drugs in high doses (psilocybin > 2 grams of dried mushrooms, lysergic acid diethylamide [LSD] > 200 micrograms) within the prior 3 months (microdosing will not require exclusion but participants would have to agree to discontinue microdosing 1 month before study entry)
* Use of tramadol, due to the potential for serotonin syndrome with concomitant use of psilocybin
* Individuals who are on MAOI (monoamine oxidase inhibitors) or who have a known sensitivity to the drug or its metabolites. Psilocybin is contraindicated in medications that are known UDP-glucuronosyltransferase (UGT) enzyme modulators
* Baseline prolongation of QT/corrected QT (QTc) interval (e.g., demonstration on a 12-lead electrocardiogram [ECG] of a QTc interval > 450 milliseconds [ms])
* A history of additional risk factors for Torsade de Points (including but not limited to: heart failure, hypokalemia, family history of Long QT Syndrome)
* The use of concomitant medications that prolong the QT/QTc interval
* Any history of cardiovascular disease such as history of myocardial infarction or congestive heart failure or cardiac arrhythmia
* The use of concomitant medications that prolong the QT/QTc interval.
* Concomitant use of efavirenz (an antiviral) which cannot be tapered
* Concomitant use of serotonin-acting supplements due to their potential for interaction with psilocybin, including 5-HTP, St John's Wort, and 'brain food' supplements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Occurrence of any adverse event graded Severe on the Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Symptoms of Anxiety and Depression assessed via the Hospital Anxiety and Depression Scale (HADS): Change in Mean Total score | At day -14, 1 week, 1 month, 2 months, 3 months, 6 months
  Measured using the Hospital Anxiety and Depression Scale (HADS). Scores range from 0 (better) to 42 (worse).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Back, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No